CLINICAL TRIAL: NCT07090928
Title: Effectiveness of Per-Operative Bupivicaine in Reducing Postoperative Pain at Port Site and Improving Mobility in Knee Arthoscopic Procedures
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Zeeshan Arif, Trainee Medical Officer, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 476/DME/KMC
Record Dates: First submitted 2025-07-04; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-06

CONDITIONS: Arthroscopic Surgery
Keywords: Bupivacaine; Postoperative Pain; Port Site Pain; Arthroscopy; Mobility Improvement; Local Anesthetic; Perioperative Analgesia; Minimally Invasive Surgery; Randomized Controlled Trial
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): group A (intervention group) will receive 5 ml of 0.5% bupivacaine infiltrated at each port site
  Interventions: Drug: 5 ml of 0.5% bupivacaine infiltrated at each port site
- Control group (Placebo Comparator): Group B (intervention group) will receive 5 ml of 0.9% Normal Saline infiltrated at each port site
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 5 ml of 0.5% bupivacaine infiltrated at each port site — 5 ml of 0.5% bupivacaine infiltrated at each port site after the arthroscopic procedures
  Arms: Intervention group
Drug: Placebo — 5ml 0.9%normal saline infiltrated at port site
  Arms: Control group

SUMMARY:
The investigator's aim is to evaluate the effectiveness of per-operative bupivacaine infiltration at arthroscopic port sites in reducing post-operative pain compared to placebo in patients undergoing knee arthroscopic procedures.

DETAILED DESCRIPTION:
Knee arthroscopy is a minimally invasive surgical procedure widely used to diagnose and treat various knee conditions such as trauma leading to meniscal tears or ligament, patellar dislocations and post-knee arthroplasty complications. Despite its less invasive nature compared to open surgery, patients often experience postoperative pain, particularly at port sites where surgical instruments are introduced which can impair early mobilization and delay recovery, and affect patient satisfaction with the procedure.

Pain management after knee arthroscopy remains a challenge in orthopaedic practice. While various analgesic strategies have been employed, including oral analgesics such as NSAIDs or opioid, intravenous analgesics or intra-articular injections. Yet, the optimal approach in managing port site pain specifically has not been fully established. Port site pain can be troublesome as it may restrict movement and contribute to delayed functional recovery after arthroscopic procedures.

Bupivacaine, a long-acting amide local anesthetic, has been used as postoperative analgesia for many procedures. Its infiltration around surgical incisions has shown promise in reducing pain after different types of surgeries. In knee arthroscopy, bupivacaine has been used intra-articularly with varying reports of its efficacy, but less attention has been given to its specific use for port site pain control and its subsequent impact on early mobility.

Recent studies have demonstrated the potential outcomes of infiltration of local anesthesia at port sites in laparoscopic procedures, suggesting similar techniques could give successful results in arthroscopic knee surgery. The effectiveness of peri-articular infiltration has been documented in total knee arthroplasty, but evidence specifically addressing arthroscopic port sites remains limited. However, a randomized controlled trial, intra-articular levo-bupivacaine demonstrated significantly lower postoperative visual analogue scale (VAS) pain scores of mean 3.2 ± 1.1 compared to bupivacaine mean VAS pain score 4.5 ± 1.3, indicating superior analgesic effect following knee arthroscopy.

This study aims to evaluate the effectiveness of per-operative bupivacaine infiltration at arthroscopic port sites in reducing postoperative pain and improving early mobility following knee arthroscopic procedures. By precisely targeting port site pain, the investigator can postulate that patients will experience greater comfort, require fewer analgesics, and achieve earlier recovery. The findings could provide valuable evidence to establish protocols for port site pain management in knee arthroscopy, potentially improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria Either Male or Female Age range: 18-70 Years Patients scheduled to undergo elective knee arthroscopic procedures Able to understand the VAS pain scale Exclusion Criteria Either Male or Female Age range: 18-70 Years Patients scheduled to undergo elective knee arthroscopic procedures Able to understand the VAS pain scale Known hypersensitivity or allergy to bupivacaine or any local anesthetics Chronic pain conditions requiring regular pain medications History of drug abuse (mainly to opioids) Pregnant women Pre-existing impaired knee mobility No willing to participate in trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Port Site Pain Score | 6 hours, 12 hours, and 24 hours postoperatively
  Pain will be measured using the Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst pain), at the port site following knee arthroscopy.

SECONDARY OUTCOMES:
Proportion of Patients Achieving Early Mobility | Assessed after 6 hours of completion of procedure
  Early mobility is defined as the ability to perform prescribed physical therapy exercises and ambulate (with assistance from a caregiver or ambulatory aids) within 6 hours after knee arthroscopic surgery. This will be recorded as a binary outcome (Yes/No) based on physiotherapist evaluation